CLINICAL TRIAL: NCT05915221
Title: Effect of SMS Reminder Use on Postoperative Respiratory and Cough Exercise Compliance of Patients After Lung Cancer Surgery
Brief Title: Effect of SMS Use on Postoperative Respiratory and Cough Exercise Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeynep Kızılcık Ozkan, Assistant professoR, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/526
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Cancer; Surgery
Keywords: short message service; breathing and coughing exercises; pulmonary lobectomy
MeSH Terms: conditions — Lung Neoplasms; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: The group that received SMS was selected as the intervention group. Patients in the control group did not receive any SMS within the scope of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group was chosen to be the group that did not receive SMS.
- SMS group (Experimental): The intervention group was chosen to be the group that received SMS messages.
  Interventions: Procedure: SMS

INTERVENTIONS:
Procedure: SMS — Receive SMS
  Arms: SMS group

SUMMARY:
Aim: This randomized controlled trial study aimed to evaluate the effect of SMS use on compliance with postoperative breathing and coughing exercises and patient satisfaction in patients undergoing pulmonary lobectomy for lung cancer surgery.

Material and methods: In the study, 62 patients who underwent lobectomy in a university hospital's thoracic surgery clinic between 01.02.2022 and 03.04.2023. The intervention group was chosen to be the group that received SMS messages.

DETAILED DESCRIPTION:
Background: Patients undergoing lung resection should be encouraged to cough, take deep breaths for pulmonary rehabilitation within the scope of enhanced recovery after surgery protocols. The success of protocols is related to patient compliance. SMS-based interventions increase compliance with medications and protocols in surgical patients and reduce hospital readmission rates, while improving patients' clinical participation and satisfaction.

Aim: This randomized controlled trial study aimed to evaluate the effect of SMS use on compliance with postoperative breathing and coughing exercises and patient satisfaction in patients undergoing pulmonary lobectomy for lung cancer surgery.

Material and methods: In the study, 62 patients who underwent lobectomy in a university hospital's thoracic surgery clinic between 01.02.2022 and 03.04.2023. The intervention group was chosen to be the group that received SMS messages.

"The Information Form", "Postoperative exercise follow-up chart", "Postoperative patient evaluation form" and "Patient satisfaction form were used in data collection. Independent sample t-test, Pearson chi- square and Mann Whitney U test were conducted for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective pulmonary lobectomy,
* having preoperative normal lung capacity (pulmonary function test result FEV1/FVC >70%),
* being compatible with the use of triflow, undergoing pulmonary lobectomy for the first time,
* volunteering to participate in the study,
* having mental competence,
* not having Turkish communication problems,
* having a personal mobile phone and accepting to send SMS,
* being an adult (≥18)

Exclusion Criteria:

* If any SMSs are not received during the study period, the patient will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
primary outcome measure | change from after implamentation 1st and 4rd days of operation.
  The primary point of the study was defined as evaluating the effect of sending SMSs, on compliance with postoperative breathing and coughing exercises undergoing pulmonary lobectomy surgery.A postoperative exercise follow-up chart includes the breathing, coughing, triflow exercises performed by the patients on the 1st and 4th postoperative days and the hours of the exercises. The mean number of breathing and coughing exercises on the first and fourth postoperative days was recorded.

SECONDARY OUTCOMES:
secondary outcome measure | change from after implamentation 4rd days of operation.
  The second point of the study was defined as evaluating the effect of sending SMSs, on patient satisfaction undergoing pulmonary lobectomy surgery. "Patient satisfaction form" were used for data collection.The patient satisfaction form" consisted of two questions. The first question questioned the satisfaction with SMS reminders. Satisfaction levels were categorized in 4 ways. Level of "very satisfied" and "satisfied" were accepted as high satisfaction level, "was not satisfied" and "was not satisfied at all" were accepted as low level.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Trakya University, Edirne
  - Turkey, Trakya University, Edirne

IPD SHARING:
Plan to Share IPD: No